CLINICAL TRIAL: NCT07387458
Title: Perception, Attitude, and Clinical Practice of Bone Turnover Markers and Vitamin D Among Health Professionals in Taiwan
Brief Title: Bone Turnover Markers and Vitamin D Survey Among Health Professionals in Taiwan
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Hsing Wu, Professor, National Cheng-Kung University Hospital
Other Study IDs: BTM & vit D survey
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Bone Remodeling; Vitamin D

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — calcium, phosphate, albumin, creatinine (Cr), alanine aminotransferase (ALT), alkaline phosphatase (ALP), and serum 25-hydroxyvitamin D [25(OH)D], iPTH, CTX, osteocalcin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals: Healthcare professionals participating in osteoporosis-related courses

SUMMARY:
This study will provide the first national overview of BTM and vitamin D utilization among healthcare professionals in Taiwan. The findings are expected to inform educational strategies, optimize clinical implementation, and support evidence-based policy development for osteoporosis management.

DETAILED DESCRIPTION:
Due to socioeconomic progress and improved healthcare, the human lifespan has increased, leading to rapid population aging and making age-related problems such as osteoporosis increasingly prominent. According to Taiwan's 2005-2008 National Nutrition Survey, the prevalence of osteoporosis among people aged 50 and older was 38.3% among women and 23.9% among men. Older adults with osteoporosis who suffer hip fractures often experience a high mortality rate. Data from Taiwan's National Health Insurance Administration shows that the one-year mortality rate for older men with hip fractures is 22%, and for women it is 15%, significantly higher than the average mortality rate for the same age group. Those who survive often require long-term care due to their inability to live independently and frequently experience refractures, further increasing the caregiving burden. Early diagnosis and appropriate intervention can prevent fractures, increasing survival time and quality of life.

Bone turnover markers (BTMs) are metabolites produced during bone formation and bone resorption. Previous studies have shown that BTMs can help predict fracture risk, assess patient adherence to medical advice, and monitor the effectiveness of drug treatment. BTMs can be divided into bone formation markers (BTMs) and bone resorption markers (BRMs). The International Osteoporosis Foundation (IOF), the International Society for Clinical Densitometry (ISCD), and the Taiwanese Osteoporosis Association (TOA) recommend that osteocalcin, bone-specific alkaline phosphatase, and procollagen type 1 amino-terminal propeptide (P1NP) be used clinically for bone formation markers. C-terminal telopeptide of type 1 collagen (CTX) and N-terminal telopeptide of type 1 collagen (NTX) can be used for bone resorption markers. Therefore, in 2021, the TOA, together with other international experts, published "Consensus statement on the use of bone turnover markers for short-term monitoring of osteoporosis treatment in the Asia-Pacific region". This statement aims to provide a reference for short-term monitoring of osteoporosis treatment efficacy and patient medication adherence, as well as for predicting future fracture risk.

Previous studies have shown that only 10% of physicians practicing in hospitals and 8% practicing in primary care use bone turnover markers (BTMs) for the diagnosis and treatment of osteoporosis; only 6.2% of patients hospitalized for fractures are advised to use BTMs for the diagnosis and treatment of osteoporosis. There is limited literature on the current clinical application of BTMs.

Therefore, this study surveyed all medical professionals attending osteoporosis-related conferences using a structured questionnaire to examine their awareness, attitudes, and current clinical use of bone turnover markers in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

- Healthcare professionals participating in osteoporosis-related courses

Exclusion Criteria:

* Diseases that may affect bone metabolism, such as cancer, stroke, or mobility impairment
* Use of medications that significantly affect bone metabolism, such as selective estrogen receptor modulators, bisphosphonates, denosumab, anabolic agents, or estrogen

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals participating in osteoporosis-related courses
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Bone formation marker | The enrollment day
  Bone formation marker concentration
Vitamin D | The enrollment day
  Vitamin D concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwanese Osteoporosis Association, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No